CLINICAL TRIAL: NCT06090045
Title: Spectrum Of Airway Involvement In Inflammatory Bowel Disease
Brief Title: Airway Involvement In Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Lecture, Assiut University
Other Study IDs: IBD&Airway
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To estimate prevalence of subclinical airway injuries among IBD patients. To investigate relationship between activity of IBD and airways

DETAILED DESCRIPTION:
Airway diseases are the most commonly described lung manifestations of inflammatory bowel disease (IBD). However, the similarities in disease pathogenesis and the sharing of important environmental risk factors and genetic susceptibility suggest that there is a complex interplay between IBD and airway diseases.Extraintestinal manifestations (EIM) commonly occur in inflammatory bowel diseases (IBD), with a prevalence rate between 21%-41% reported in various series. Crohn's disease (CD) presents with EIM more frequently than ulcerative colitis (UC). Pulmonary involvement complicating IBD was originally considered rare (with a frequency rate < 1%), but the first case series published in 1976 assisted in better recognition, evaluation and description of IBD related respiratory disease. Pulmonary involvement is often asymptomatic and may be detected solely on the basis of abnormal screening tests. This review will focus on the involvement of the airways in the context of IBD. Although IBD related PM were originally considered rare, certain population-based studies have revealed significant interrelationships between the lungs and IBD. Bernstein and colleagues in a large population-based study in North America in 2005 reported that airway disorders in general (including asthma and bronchitis) were the most common extraintestinal manifestation in subjects with CD and the second most common in subjects with UC, with the prevalence of asthma in this population between 7%-8%. In another retrospective study from the opposite view, Birring reported that IBD was 4 times more prevalent among patients with airway diseases, particularly non-asthmatic patients with productive cough, than in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Patients attended to IBD clinic at Tropical Department

Exclusion Criteria:

1. Age: less than 18 years
2. Unstable patients or need for ICU admission

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After taking the informed consent, full history will be taken from all patients participating in the study. Detailed clinical examination and routine laboratory investigations (complete blood count, liver function test, urea, creatinine and ESR) will be done Clinical notes will be obtain and review for all patients with a diagnosis of IBD (history of bowel surgery (for IBD, or indication not stated), use of 5-aminosalicylates or immunomodulators (if indication not stated) ).
  Diagnosis of IBD will confirm on the basis of a consistent clinical picture with endoscopic and histological confirmation, or characteristic radiological appearances.
  Airways disease will classify on the following grounds: asthma,.COPD:,Bronchiectasis,.Chronic bronchitis:
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Predictors of airway diseases in patients with IBD | baseline
  FROM risk factors

SECONDARY OUTCOMES:
-Prevalence of of subclinical airway injuries among IBD patients presented to Tropical Department in Assiut University Hospital | baseline
  from statistical anyalasis

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Salama, MD, Study Chair — Assiut University

REFERENCES:
- [Background] Vutcovici M, Brassard P, Bitton A. Inflammatory bowel disease and airway diseases. World J Gastroenterol. 2016 Sep 14;22(34):7735-41. doi: 10.3748/wjg.v22.i34.7735. PMID 27678355
- [Background] Byrd KM, Gulati AS. The "Gum-Gut" Axis in Inflammatory Bowel Diseases: A Hypothesis-Driven Review of Associations and Advances. Front Immunol. 2021 Feb 19;12:620124. doi: 10.3389/fimmu.2021.620124. eCollection 2021. PMID 33679761